CLINICAL TRIAL: NCT05391737
Title: Cardiac Function in Swimming-Induced Pulmonary Edema (SIPE) - a Case Control Study
Brief Title: Cardiac Function in Swimming-Induced Pulmonary Edema (SIPE)
Status: Recruiting | Type: Observational
Sponsor: Dalarna County Council, Sweden (Other)
Responsible Party: Principal Investigator, Maria Hårdstedt, Dr. Maria Hårdstedt, PhD, Specialist Internal Medicine, Dalarna County Council, Sweden
Other Study IDs: SIPE Cardiac function 001
Record Dates: First submitted 2022-05-17; First posted 2022-05-26 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Swimming Induced Pulmonary Edema (SIPE); Pulmonary Edema; Lung Diseases; Heart Function Tests
Keywords: Echocardiography; Electrocardiography; Troponin
MeSH Terms: conditions — Pulmonary Edema; Lung Diseases | interventions — Echocardiography; Electrocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- patients with SIPE: Adult patients (age ≥18 years) with SIPE-diagnosis during "Vansbrosimningen" and peripheral oxygen saturation ≤95%. SIPE-diagnosis based on pulmonary edema on lung ultrasound.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Electrocardiogram (ECG); Diagnostic Test: Cardiac biomarkers
- control group: Swimmers completing "Vansbrosimningen" without respiratory symptoms or signs of pulmonary edema on lung ultrasound. Matched to patients with SIPE for age and gender.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Electrocardiogram (ECG); Diagnostic Test: Cardiac biomarkers

INTERVENTIONS:
Diagnostic Test: Echocardiography — Echocardiography after swimming (acute) and at rest (baseline)
Diagnostic Test: Electrocardiogram (ECG) — Electrocardiogram (ECG) after swimming (acute) and at rest (baseline)
Diagnostic Test: Cardiac biomarkers — high sensitive (hs)-Troponin I and N-terminal pro-brain natriuretic peptide (NT-pro-BNP) after swimming (acute) and at rest (baseline)

SUMMARY:
Acute or chronic cardiac dysfunction could be a contributing factor to swimming-induced pulmonary edema (SIPE). Knowledge on cardiac function in SIPE is limited and recommendations for cardiac evaluation of patients with SIPE are lacking. The present study was designed to assess cardiac function in patients with SIPE and in asymptomatic swimmers.

DETAILED DESCRIPTION:
Swimming induced pulmonary edema (SIPE) is an unusual condition occuring during swimming in cold open water. SIPE is characterized by acute onset of dyspnea and cough, excessive sputum and occasionally hemoptysis. Reversible myocardial dysfunction has been described in swimmers with SIPE and divers with immersion pulmonary edema (IPE). Cardiac dysfunction has also been discussed as a contributing factor triggering SIPE. However, prevalence, severity and prognosis of myocardial dysfunction in patients with SIPE is unknown. Official recommendations for cardiac evaluation of patients after an acute episode of SIPE is lacking.

This case-control-study intends to assess cardiac function in patients with SIPE and in asymptomatic swimmers. We study a large cohort of approximately 12 000 swimmers during Vansbrosimningen, Sweden's biggest annual open water event, with a yearly incidence of SIPE of about 0,4%. Cardiac function is evaluated after swimming as well as at rest by echocardiography, 12-lead electrocardiogram and cardiac biomarkers (Troponin I, NT-pro-BNP).

ELIGIBILITY:
Inclusion Criteria:

for patients:

* respiratory symptoms during or after swimming at the Vansbrosimningen open water swimming event
* diagnosis SIPE by signs of pulmonary edema on lung ultrasound
* peripheral oxygen saturation ≤95%

for controls:

* completion of a swimming race of the Vansbrosimningen open water swimming event.
* no respiratory symptoms during or after swimming
* no signs of pulmonary edema on lung ultrasound
* matched to patients with SIPE regarding sex and age

Exclusion criteria:

* declined consent
* hemodynamic instability or decreased consciousness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adults (age ≥18 years) that participate in a swimming race during Vansbrosimningen open water swimming event.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Acute Echocardiography | within 4 hours after termination of swimming
  Transthoracic echocardiography with parasternal, apical and subcostal views. Including measurement of ventricular wall size, left ventricular strain, ejection fraction according to the modified Simpson method, diastolic function (using tissue doppler, mitral flow and pulmonary vein flow), right ventricular tricuspid annular plane systolic excursion (TAPSE), pressure gradient over the tricuspid valve, assessment of valve dysfunction, size and respiratory variation of the inferior vena cava, assessment of pericardial fluid.
Acute Electrocardiogram (ECG) - Rytm analysis | within 4 hours after termination of swimming
  12-lead electrocardiogram (ECG). Rytm analysis and frequency (beats per minute)
Acute Electrocardiogram (ECG) - Heart axis | within 4 hours after termination of swimming
  12-lead electrocardiogram (ECG). Assessment of QRS-axis (degrees)
Acute Electrocardiogram (ECG) - Amplitudes and intervals | within 4 hours after termination of swimming
  12-lead electrocardiogram (ECG). Duration of PQ-interval (ms), QRS-complex (ms), QT-interval (ms), QRS amplitude (mV)
Acute Electrocardiogram (ECG) - Signs of myocardial ischemia | within 4 hours after termination of swimming
  12-lead electrocardiogram (ECG). ST-elevation, ST-depression, T-wave inversion, Q wave.
Acute cardiac biomarkers - Troponin I | 4-6 hours after termination of swimming
  Venous samples. Measurement of hs-Troponin I (ng/L).
Acute cardiac biomarkers - NT-pro-BNP | 4-6 hours after termination of swimming
  Venous samples. Measurement of NT-pro-BNP (ng/L)

SECONDARY OUTCOMES:
Baseline Echocardiography | within 12 months after swimming
  Transthoracic echocardiography with parasternal, apical and subcostal views. Examination at rest. Including measurement of ventricular wall size, left ventricular strain, ejection fraction according to the modified Simpson method, diastolic function (using tissue doppler, mitral flow and pulmonary vein flow), right ventricular tricuspid annular plane systolic excursion (TAPSE), pressure gradient over the tricuspid valve, assessment of valve dysfunction, size and respiratory variation of the inferior vena cava, assessment of pericardial fluid.
Baseline Electrocardiogram (ECG) - Rytm analysis | within 12 months after swimming
  12-lead Electrocardiogram (ECG). Examination at rest. Rytm analysis and frequency (beats per minute)
Baseline Electrocardiogram (ECG)- Heart axis | within 12 months after swimming
  12-lead Electrocardiogram (ECG). Examination at rest. Assessment of QRS-axis (degrees)
Baseline Electrocardiogram (ECG) - Amplitudes and intervals | within 12 months after swimming
  12-lead Electrocardiogram (ECG). Examination at rest. Duration of PQ-interval (ms), QRS-complex (ms), QT-interval (ms), QRS amplitude (mV)
Baseline Electrocardiogram (ECG) - Signs of myocardial ischemia | within 12 months after swimming
  12-lead Electrocardiogram (ECG). Examination at rest. ST-elevation, ST-depression, T-wave inversion, Q wave.
Baseline cardiac biomarkers - Troponin I | within 12 months after swimming
  Venous samples. Measurement of hs-Troponin I (ng/L). Examination at rest
Baseline cardiac biomarkers - NT-pro-BNP | within 12 months after swimming
  Venous samples. Measurement of NT-pro-BNP (ng/L). Examination at rest

CONTACTS AND LOCATIONS:
Locations (1):
- Center of Clinical Research Dalarna, Falun, Sweden

IPD SHARING:
Plan to Share IPD: No